CLINICAL TRIAL: NCT00618566
Title: A Peer Implemented Cognitive Behavioral Group Therapy Intervention for Use With Women With Physical Disabilities With Secondary Depression
Brief Title: Group Therapy Program for Women With Physical Disabilities
Acronym: CBT-WPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dena Hassouneh, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDRR; H133G060135
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Depressive Symptoms
Keywords: Women with physical Disabilities; Secondary Conditions; Depression; Cognitive Behavioral Therapy; Consumer Control
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oregon (Experimental)
  Interventions: Behavioral: WPD and Depression Treatment Group

INTERVENTIONS:
Behavioral: WPD and Depression Treatment Group — Intervention selected will depend on Phase I data analysis.

SUMMARY:
More women with disabilities (30%) report "feelings such as sadness, unhappiness, or depression that prevent them from being active" compared to women without disabilities (8%). The contexts of the lives of WPD, which often include high rates of poverty, architectural and attitudinal barriers, and higher vulnerability to violence and abuse, contribute to this mental health disparity. To help address this disparity, the overall goals of this pilot study are to: 1)1. Develop a cognitive behavioral group therapy intervention to address the specific needs of WPD who experience depressive symptoms; and 2. Pilot-test the intervention to preliminarily evaluate its efficacy using a mixed-methods approach. The proposed and revised study outcomes were derived from our previous work with WPD as well as from feedback obtained from community meetings conducted since our last submission of this proposal. A pilot of the modified intervention with a total of 90 participants will be conducted using a using a wait list control design. The decision to use a wait list control design was made jointly with our community partners to ensure that all WPD participating in the study have access to the intervention.

DETAILED DESCRIPTION:
The project will use a longitudinal mixed method research design. Phase I will utilize focus groups conducted with WPD to support development of the group therapy program. Phase II will evaluate the efficacy of the intervention using a randomized design. Measures to protect human subjects include development of detailed safety and referral protocols including 24 hour access to emergency mental health assessment and intervention as needed.

ELIGIBILITY:
Inclusion Criteria:

* Women with physical disabilities age 18 and older who require some form of accommodation and experience significant depressive symptoms as defined by a cut off score of 16 or greater on the CES-D.

Exclusion Criteria:

* Women currently receiving other psychotherapy treatment
* Women who are psychotic or have significant cognitive impairment
* Women who are actively suicidal with intent and plan
* Women who have discontinued or initiated antidepressant medications within an 4 week time period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2007-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The following hypothesis is specific to the primary outcome: Hypotheses: 1. WPD receiving the intervention will demonstrate a greater improvement in depressive symptom scores compared to participants in the wait-list control groups. | 3 years

SECONDARY OUTCOMES:
Secondary Outcomes: Hypothesis 2: the intervention group will demonstrate a greater improvement in coping and problem-solving skills, health behavior, body image and sexual self-esteem and loneliness compared to wait-listed controls. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dena Hassouneh, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States